CLINICAL TRIAL: NCT03722576
Title: Investigation of the Activity of Vidofludimus Calcium, a Novel, Orally Available, Small Molecule Inhibitor of Dihydroorotate Dehydrogenase, as a Treatment for Primary Sclerosing Cholangitis (PSC)
Brief Title: Vidofludimus Calcium for Primary Sclerosing Cholangitis
Acronym: PSC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Elizabeth Carey (Other)
Collaborators: Arizona State University (Other)
Responsible Party: Sponsor-Investigator, Elizabeth Carey, Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IND140679
Record Dates: First submitted 2018-10-25; First posted 2018-10-29 (Actual); Results first posted 2021-06-02 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Primary Sclerosing Cholangitis
MeSH Terms: conditions — Cholangitis, Sclerosing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vidofludimus Calcium (VC) (Experimental): Daily dosing of VC over 6 months
  Interventions: Drug: Vidofludimus calcium

INTERVENTIONS:
Drug: Vidofludimus calcium — During the 6-month treatment period, subjects will receive 30 mg VC orally once daily. This will be preceded by a lead-in dosing period where subjects will receive 15 mg VC once daily for 1 week.
  Other Names: IMU-838

SUMMARY:
To examine the safety, tolerability, and efficacy of daily dosing with vidofludimus calcium over a 6-month period.

DETAILED DESCRIPTION:
Investigators will assess the following:

1. Changes on serum alkaline phosphatase levels at 3 & 6 months.
2. Changes in other liver biochemistries at 3 & 6 months.
3. Changes in IL-17 &IFNγ levels at 6 weeks and 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject age 18-75 years
2. Diagnosis of PSC consistent with the guidelines published by the AASLD. All subjects must have an elevated serum ALP of at least 1.5 times upper limit of normal (ULN) at baseline plus cholangiographic evidence of PSC (MRI, endoscopic retrograde cholangiography, or direct cholangiography).
3. Indirect bilirubin <1.2 times the ULN
4. An ultrasound (or equivalent imaging modality) that excludes biliary obstruction and malignancy within 6 months of study enrollment
5. PSC with or without inflammatory bowel disease, such as ulcerative colitis or Crohn's disease
6. Must agree to comply with the study protocol and provide informed consent

Exclusion Criteria:

1. Pregnancy, attempting to become pregnant, or breastfeeding
2. Active hepatitis A or B infection
3. Active hepatitis C infection (antibody positive); patients with a history of hepatitis C infection will be eligible for this study if they have undetectable levels of HCV RNA
4. HIV/AIDS (per medical record or HIVAb/HIA antigen), tuberculosis, or positive interferon-gamma assay (IGRAs) for Mycobacterium tuberculosis
5. Other cholestatic liver disease such as primary biliary cholangitis and cholestatic diseases of pregnancy
6. Metabolic liver diseases such as Wilson's disease, Gilbert's syndrome or hemochromatosis
7. Serum uric acid levels at screening >1.2 ULN
8. Inherited diseases of the liver such as α-1 antitrypsin deficiency
9. Immunoglobulin G4-related cholangitis
10. PSC with concomitant autoimmune hepatitis (AIH) and/or primary biliary cholangitis
11. Secondary sclerosing cholangitis (SSC)
12. Active acute ascending cholangitis requiring antibiotics
13. CCA (malignant biliary stricture, neoplasm, and cytology/histopathology or positive fluorescence in situ hybridization (FISH) consistent with adenocarcinoma of the bile duct)
14. A liver biopsy, if one has been previously obtained, which showed non-alcoholic steatohepatitis (NASH). Patients with suspected fatty liver by imaging will not be excluded.
15. Presence of complications of advanced PSC such as hepatic encephalopathy, portal hypertension, hepato-renal syndrome, and hepato-pulmonary syndrome
16. History of liver transplantation, anticipated need for liver transplantation within 12 months from randomization, a Model of End-stage Liver Disease (MELD) score of ≥15, or a Child Pugh score >6
17. Ongoing alcohol abuse (>4 drinks per day for men, and >2 drinks per day for women)
18. Moderate-to-severe renal impairment with a calculated creatinine clearance of <60mL/min
19. Any other conditions or abnormalities that, in the opinion of the investigator, may compromise the safety of the subject or interfere with the subject participating in or completing the study
20. Evidence of, or treatment for, C. difficile infection within 30 days before the initiation of the study drug
21. Evidence of active C. difficile infection during the screening phase confirmed by a positive C. difficile toxin B
22. Subjects who have been treated for intestinal pathogens other than C. difficile infection within 30 days prior to study drug initiation
23. Received or plan to receive live vaccine within 30 days prior to, and through the end of the study
24. Use of methotrexate at dose ≥17.5mg/week
25. Rosuvastatin exceeding 10 mg daily

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Carey, MD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Phoenix, Arizona
  - Arizona State University, Tempe, Arizona
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Vidofludimus Calcium (VC): Daily dosing of Vidofludimus Calcium (VC) over 6 months
  Vidofludimus calcium: During the 6-month treatment period, subjects received 30 mg VC orally once daily. This was preceded by a lead-in dosing period where subjects received 15 mg VC once daily for 1 week.
Period: Overall Study
Arm/Group | Vidofludimus Calcium (VC)
Started | 18
Completed | 11
Not Completed | 7
Not completed — Withdrawal by Subject | 3
Not completed — Adverse Event | 2
Not completed — Physician Decision | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Vidofludimus Calcium (VC): Daily dosing of VC over 6 months
  Vidofludimus calcium: During the 6-month treatment period, subjects received 30 mg VC orally once daily. This was preceded by a lead-in dosing period where subjects received 15 mg VC once daily for 1 week.
Arm/Group | Vidofludimus Calcium (VC)
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.7 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 18
  Not Hispanic or Latino | 17
  Hispanic or Latino | 1
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Subjects Who Experience a Positive Outcome as Measured by Combination of Serum Alkaline Phosphatase (ALP) and Aspartate Aminotransferase (AST) Levels.
Description: The number of subjects who have both an ALP reduction from baseline to week 24 that is greater or equal to 25% and their AST increase from baseline is less than or equal to 33% at week 24. ALP measured as international units per liter (IU/L). AST measured as international units per liter (IU/L).
Time Frame: Baseline to 24 weeks
Population: Only subjects who completed treatment were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Vidofludimus Calcium (VC)
Number analyzed (Participants) | 11
Participants | 3

2. Secondary Outcome: Abnormal Aspartate Aminotransferase (AST)
Description: Number of subjects with abnormal (not within normal range) AST levels. AST is an enzyme found in high amounts in liver, heart, and muscle cells. This test is mainly done along with other tests such as alkaline phosphatase and bilirubin to diagnose and monitor liver disease. This test evaluates hepatocyte integrity, as serum levels of this enzyme rise in response to a variety of forms of injury to hepatic cells. The normal range is 5 to 40 U/L . Units: U/L
Time Frame: Baseline to 24 weeks
Population: Only subjects who completed the lab tests at 24 weeks were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Vidofludimus Calcium (VC)
Number analyzed (Participants) | 10
Participants | 8

3. Secondary Outcome: Abnormal Alanine Aminotransferase (ALT)
Description: Number of subjects with abnormal (not within normal range) ALT levels. An enzyme normally present in liver and heart cells that is released into the bloodstream when the liver or heart is damaged. The blood ALT levels are elevated with liver damage (for example, from viral hepatitis) or with an insult to the heart (for example, from a heart attack). The normal range is 7 to 56 U/L. Units: U/L
Time Frame: 24 weeks
Population: Only subjects who completed the lab tests at 24 weeks were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Vidofludimus Calcium (VC)
Number analyzed (Participants) | 10
Participants | 8

4. Secondary Outcome: Abnormal Total Bilirubin
Description: Number of subjects with abnormal (not within normal range) Total Bilirubin levels. Bilirubin is a yellowish pigment found in bile, a fluid made by the liver. A small amount of older red blood cells are replaced by new blood cells every day. Bilirubin is left after these older blood cells are removed. The liver helps break down bilirubin so that it can be removed from the body in the stool. The normal range for total bilirubin is 0.3 to 1.2 mg/dL Units: mg/dL
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Vidofludimus Calcium (VC)
Number analyzed (Participants) | 10
Participants | 3

5. Secondary Outcome: Abnormal Direct Bilirubin
Description: Number of subjects with abnormal (not within normal range) direct bilirubin levels. In the liver, bilirubin is changed into a form that your body can get rid of. This is called conjugated bilirubin or direct bilirubin. This bilirubin travels from the liver into the small intestine. A very small amount passes into your kidneys and is excreted in your urine. Normal range for direct bilirubin is 0.3 and 1.2 milligrams per deciliter (mg/dL). Units: mg/dL
Time Frame: 24 weeks
Population: Only subjects who completed the lab tests at 24 weeks were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Vidofludimus Calcium (VC)
Number analyzed (Participants) | 10
Participants | 4

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline to end of study, approximately 8 months
Arm/Group | Vidofludimus Calcium (VC)
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 12/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vidofludimus Calcium (VC) (N=18)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Alkaline phosphatase increase (Investigations) | 1 (1)
Allergic reaction (Immune system disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Fatigue (General disorders) | 1 (1)
Fever Pyrexia (General disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1)
Achy neck and shoulders (Musculoskeletal and connective tissue disorders) | 1 (1)
Bleeding from ileostomy (Gastrointestinal disorders) | 1 (1)
Cold (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Discolored Stool (Gastrointestinal disorders) | 1 (1)
Flu (General disorders) | 1 (1)
Gatroenteritis (Gastrointestinal disorders) | 1 (1)
Lipoma on back (Skin and subcutaneous tissue disorders) | 1 (1)
Miscarriage (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Upper right abdominal pain (Gastrointestinal disorders) | 1 (1)
Worsened loose stools (Gastrointestinal disorders) | 1 (1)
Worsening liver enzymes (Investigations) | 1 (1)
Cholangitis (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-23): https://cdn.clinicaltrials.gov/large-docs/76/NCT03722576/Prot_SAP_000.pdf